CLINICAL TRIAL: NCT03197220
Title: The Impact of Fish and Walnut Consumption on Cardiovascular Risk Factors in Overweight and Obese Females: A Randomized Clinical Trial
Brief Title: Omega-3 and Cardiovascular Risk Factors and Kidney Related Biomarkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Leila Azadbakht, Professor, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: omega-3
Record Dates: First submitted 2017-03-03; First posted 2017-06-23 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2017-03

CONDITIONS: Cardiovascular Risk Factor and Kidney Related Biomarkers
MeSH Terms: interventions — In Situ Hybridization, Fluorescence; PR-10 protein, walnut birch pollen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- fish (Experimental)
  Interventions: Other: fish
- walnut (Experimental)
  Interventions: Other: walnut
- fish-walnut (Experimental)
  Interventions: Other: fish-walnut

INTERVENTIONS:
Other: fish — 300 gr/week fish
  Arms: fish
Other: walnut — 18 walnut per week
  Arms: walnut
Other: fish-walnut — 150 gr fish and 9 walnut per week
  Arms: fish-walnut

SUMMARY:
In this study, 99 overweight or obese women that referred to the Clinic Nutrition to lose weight were randomly divided into three groups according to body mass index (BMI) by random-number table (figure1). We attempted to match all three groups for BMI, probable medications, and age. Subjects were excluded if they had risk factors of cardiovascular diseases or allergic reactions to fish or walnut, or received lowering blood glucose or lipid profile agents. Also, participants with weak economic status could not enter to this study (due to the high cost of fish and walnuts). Before the start of this study, the information in the form of questionnaire about demographic, medical history, and medication use, was completed. Participants were aware about overview of this study, and completed the consent form. The NATIONAL INSTITUTED FOR MEDICAL RESEARCH DEVELOPMENT (NIMAD), approved all procedures involving human subjects. The study has been done in accordance with the ethical standards in declaration of Helsinki.

Then all of the three groups received a low-calorie diet in order to lose weight. The distribution of macronutrients was similar in three groups (carbohydrate 55%, fat 33%, and protein 17%). The amount of different fatty acids (saturated, unsaturated with mono double bond, and polyunsaturated fatty acids) intake in these diets was the same but the sources of omega-3 between these groups were different. In the first group, subjects were instructed to consume 300 gram fatty fish, such as Salmon fish during a week in two separated meals (each meal 150 gr fatty fish) and to avoid consumption of plant sources of omega-3 (soybean oil, canola, flaxseed and walnuts). In the second group, subjects were asked to consume walnuts three times a week and each time two walnuts (totally 18 walnuts/wk) and avoid the consumption of fish. And in the third group, subjects were recommended to consume 150 g fatty fish during a week and nine walnuts. The amount of omega-3 fatty acids considered in this study covered the typical recommended intake (0.3 to 0.5 g/d of EPA+DHA and 0.8 to 1.1 g/d of ALA)(14). Dietary intakes of all patients were controlled by a dietitian and they were followed for 12 weeks. Dietary intakes were assessed by three dietary records (one weekend and two week days).

DETAILED DESCRIPTION:
This is a clinical trial which conducted on over weight and obese female.

ELIGIBILITY:
Inclusion Criteria:

* over weight or obese

Exclusion Criteria:

* have any diseases

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — overweight or obese female that referred to the Clinic Nutrition to lose weight
Enrollment: 99 (Actual)
Dates: Start 2015-11-22 (Actual); Primary Completion 2016-11-21 (Actual); Study Completion 2017-01-20 (Actual)

PRIMARY OUTCOMES:
the change of biochemical factor levels | 12 weeks
  Systolic and diastolic blood pressures (SBP and DBP) will measured twice after 15 min of rest in sitting and comfortably position using a standard mercury sphygmomanometer. Blood sugar (FBS) will measured on the day of blood sampling and quantified by colorimetric method by the glucose oxidize technique. hs-CRP will measured by The Immunoturbidimetry method with with a polyclonal antibody (Pars Azmoon Inc). Serum concentrations of, high-density lipoprotein cholesterol(HDL-C), low-density lipoprotein cholesterol (LDL-C) and triglyceride (TG) will quantified using commercially available enzymatic reagents (Pars Azmoon, Tehran, Iran) adapted to an autoanalyzer system (Selectra E, Vitalab, Holliston, the Netherlands).

SECONDARY OUTCOMES:
height | 12 week
  meter
weight | 12 week
  kg
BUN | 12 WEEK
creatinine | 12 WEEK

OTHER OUTCOMES:
body mass index | 12 week
  BMI was calculated as body weight in kg divided by height in m2.
physical activities | 12 week
  We asked participants to record the duration of all physical activities in 24h for three days at weeks 3, 6, 9 and 12 of the intervention. Then the recorded physical activities were multiplied by the relevant metabolic equivalents task hours per day (MET-h/d) and were calculated the MET.h/d values of all activities to obtain the value of physical activity in a day.
Hs-CRP | 12 week
  Hs-CRP was measured by the Immunoturbidimetry method with a polyclonal antibody (Pars Azmoon Inc).
high-density lipoprotein cholesterol (HDL-C), LDL-C and TG | 12 week
  were quantified using commercially available enzymatic reagents (Pars Azmoon, Tehran, Iran) adapted to an autoanalyzer system (Selectra E, Vitalab, Holliston, the Netherlands).

REFERENCES:
- [Derived] Fatahi S, Haghighatdoost F, Larijani B, Azadbakht L. Effect of Weight Reduction Diets Containing Fish, Walnut or Fish plus Walnut on Cardiovascular Risk Factors in Overweight and Obese Women. Arch Iran Med. 2019 Oct 1;22(10):574-583. PMID 31679359